CLINICAL TRIAL: NCT02769247
Title: Efficacy of Intrauterine Lidocaine and Naproxen for Pain Control With Intrauterine Device Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 384645-5
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Contraception; Pain
Keywords: naproxen; lidocaine; intrauterine device; IUD; pain
MeSH Terms: conditions — Pain | interventions — Naproxen; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Experimental): Patient will receive placebo oral medication and intrauterine normal saline prior to IUD insertion
  Interventions: Drug: placebo
- Naproxen/Normal saline (Experimental): Patient will receive naproxen and intrauterine normal saline prior to IUD insertion
  Interventions: Drug: Naproxen; Drug: placebo
- Placebo oral medication/Lidocaine (Experimental): Patient will receive placebo oral medication and intrauterine lidocaine prior to IUD insertion
  Interventions: Drug: Lidocaine; Drug: placebo
- Naproxen/Lidocaine (Experimental): Patient will receive naproxen and intrauterine lidocaine prior to IUD insertion
  Interventions: Drug: Naproxen; Drug: Lidocaine

INTERVENTIONS:
Drug: Naproxen — Oral naproxen vs placebo
  Arms: Naproxen/Lidocaine; Naproxen/Normal saline
Drug: Lidocaine — Intrauterine lidocaine vs normal saline
  Arms: Naproxen/Lidocaine; Placebo oral medication/Lidocaine
Drug: placebo — either normal saline or empty oral capsule
  Arms: Naproxen/Normal saline; Placebo; Placebo oral medication/Lidocaine

SUMMARY:
To compare the efficacy of intrauterine lidocaine and oral naproxen sodium on discomfort and pain of patients undergoing intrauterine device insertion.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study with women that will be recruited from our outpatient obstetrics and gynecology clinic. Women desiring intrauterine device insertion will be invited to participate.

The investigators plan to recruit women desiring intrauterine device insertion into one of four groups: A: placebo/normal saline infusion; B: placebo/lidocaine infusion; C: Saline infusion/ naproxen; D: lidocaine infusion/ naproxen.

ELIGIBILITY:
Inclusion Criteria:

* DEERS-eligible reproductive age women (i.e. Tricare beneficiaries)
* age 18 years and older
* desiring Paragard or Mirena intrauterine device insertion

Exclusion Criteria:

* Current pregnancy
* cervical stenosis
* severe medical illness
* known allergy or sensitivity to lidocaine or naproxen
* peptic ulcer disease
* current pelvic inflammatory disease
* patients with known renal insufficiency
* patients using chronic NSAIDs or on chronic pain medication
* women desiring Skyla IUD insertion will also be excluded due to infrequency of insertions at WRNMMC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dunlow, MD, Principal Investigator — WRNMMC
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Miles SM, Shvartsman K, Dunlow S. Intrauterine lidocaine and naproxen for analgesia during intrauterine device insertion: randomized controlled trial. Contracept Reprod Med. 2019 Sep 10;4:13. doi: 10.1186/s40834-019-0094-0. eCollection 2019. PMID 31516731

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Started | 40 | 40 | 40 | 40
Completed | 38 (unable to insert IUD in one patient; 1 pt decided against study participation after enrollment) | 40 | 39 (1 took non-study med after enrollment/randomization, before IUD insertion (excluded from study)) | 39 (1 patient decided against study participation after enrollment/randomization)
Not Completed | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine | Total
Number analyzed (Participants) | 39 | 40 | 39 | 39 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 40 | 39 | 39 | 157
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 39 | 39 | 157
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 40 | 39 | 39 | 157

OUTCOME MEASURES:

1. Primary Outcome: Pain Control With IUD Insertion
Description: visual analog scale (0-10) as assessed by patient within 30 minutes after IUD insertion. Scale is from a minimum of 0, with maximum of 10 with higher scores denoting more pain
Time Frame: within 30 minutes after IUD insertion
Population: There is one patient in placebo arm that did not receive IUD due to difficulty with insertion.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 38 | 40 | 39 | 39
units on a scale | 3.606 (.372) | 3.088 (.367) | 2.83 (.372) | 3.382 (.372)

2. Secondary Outcome: Physician Perceived Pain Control During IUD Insertion
Description: visual analog scale (0-3) as assessed by physician within 30 minutes after IUD insertion Scale is from a minimum of 0, with maximum of 3 with higher scores denoting more pain
Time Frame: within 30 minutes after IUD insertion
Population: There was one patient in placebo arm unable to have her IUD placed due to difficulty with insertion. She was removed from the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 38 | 40 | 39 | 39
units on a scale | .59 (.8) | .48 (.11) | .56 (.09) | .77 (.11)

3. Secondary Outcome: Patient Satisfaction With IUD
Description: Patient satisfaction as rated on a 1-5 scale 30 days post insertion. Scale of 5 means highly satisfied, 1 means unsatisfied.
Time Frame: 30 days post insertion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 38 | 40 | 39 | 39
units on a scale | 4.423 (.16) | 4.325 (.145) | 4.264 (.153) | 4.358 (.147)

4. Secondary Outcome: Difficulty IUD Insertion
Description: as rated by the physician. Very easy/easy were rated as "easy" whereas difficult/very difficult is difficult.
Time Frame: within 30 minutes of IUD insertion
Population: Overall number of participants analyzed for placebo arm is different due to 1 of the subjects not able to have their IUD inserted due to difficulty of procedure. They were included in this analysis as an attempt had been made to insert device.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 38 | 40 | 39 | 39
Participants
  Easy | 36 | 38 | 38 | 38
  Difficult | 2 | 2 | 1 | 1

5. Secondary Outcome: Perceived Pain 30 Days Post Insertion
Description: survey patient 30 days later to determine her recollection of pain during insertion (0-10); 10 being the most pain. One patient had no IUD initially inserted and was not included; each arm had patients lost to follow up (3 in placebo arm, 2 in naproxen arm, 4 in placebo/oral medication arm).
Time Frame: 30 days post IUD insertion
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 33 | 38 | 35 | 39
units on a scale | 3.12 (.40) | 2.97 (.43) | 3.2 (.48) | 3.04 (.42)

6. Post Hoc Outcome: Paragard vs Mirena IUD
Description: difference in pain ratings during IUD insertion as assessed by visual analog scale by both patient (0-10 with 10 being the most pain, 0 no pain) within 30 minutes post insertion classified by IUD type. This measure is made to address whether type of IUD affected pain perception.
Time Frame: visual analog scale as assessed by patient and physician both within 30 minutes post insertion
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Mirena: All treatment arms that received this type IUD
- Paragard IUD: All treatment arms
Arm/Group | Mirena | Paragard IUD
Number analyzed (Participants) | 79 | 77
units on a scale | 3.02 (.25) | 3.49 (.25)

7. Post Hoc Outcome: Paragard vs Mirena IUD Pain Medication Use
Description: Patient's recall of self administered pain medication within 24 hours after IUD insertion as reported 30 days post insertion. Denoted as "yes " or "no". This measure was to assess whether any difference in pain perception between patients receiving different types of IUD.
Time Frame: 30 days post insertion
Population: These participants reflect the number of patients that were able to be successfully contacted approximately 30 days after their IUD insertion.
Measure: Count of Participants; unit: Participants
Groups:
- Mirena Medication Use: All treatment arms receiving mirena IUD
- Paragard: All treatment arms receiving paragard IUD
Arm/Group | Mirena Medication Use | Paragard
Number analyzed (Participants) | 73 | 72
Participants
  Medication used postprocedure | 16 | 23
  No medication use post procedure | 57 | 49

8. Post Hoc Outcome: Paragard IUD Medication Use 30 Day Assessment
Description: Assessment of whether patient had used analgesics in first 24 hrs after Paragard IUD insertion. Quantified yes or no.
Time Frame: 30 days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 17 | 20 | 18 | 17
Participants
  Yes, used analgesics | 7 | 4 | 5 | 7
  No medication use | 10 | 16 | 13 | 10

9. Post Hoc Outcome: Assessment of Analgesic Use in Mirena IUD Patients Within 24 Hrs When Queried at Day 30
Description: Assessment at day 30 if patients used analgesics within 24 hrs post Mirena IUD insertion
Time Frame: 30 days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
Number analyzed (Participants) | 16 | 20 | 18 | 19
Participants
  Yes, used analgesics | 5 | 5 | 3 | 3
  No analgesics used | 11 | 15 | 15 | 16

ADVERSE EVENTS:
Arm/Group | Placebo | Naproxen/Normal Saline | Placebo Oral Medication/Lidocaine | Naproxen/Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/39 | 0/39

LIMITATIONS AND CAVEATS:
Sample size is limitation. Single site conducting study using single insurance payer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No